CLINICAL TRIAL: NCT03085186
Title: Treatment With Crizotinib Single Patient Expanded Access IND 134375
Status: No longer available | Type: Expanded Access
Sponsor: Jean M. Tersak, M.D. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Jean M. Tersak, M.D., Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO17030033
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Inflammatory Myofibroblastic Tumour
MeSH Terms: conditions — Granuloma, Plasma Cell | interventions — Crizotinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Crizotinib

SUMMARY:
Two year old male with a new diagnosis of Inflammatory Myofibroblastic Tumour. The patient presented with 2 months of intermittent fever and 1-2 weeks of abdominal distention and constipation. An abdominal mass was palpable on exam and US concerning was for neoplasm of abdomen.

Treatment with Crizotinib will be utilized to reduce the size of the lesion and create more optimal tissue plains between vital structures prior to attempted surgical resection would greatly reduce potential morbidity for this patient.

ELIGIBILITY:
Inclusion Criteria:

* This treatment plan is intended for the use of Crizotinib in the treatment of a single patient with Inflammatory Myofibroblastic Tumour

Exclusion Criteria:

* Not applicable as Expanded Access only includes one patient

Ages: 2 Years to 2 Years | Sex: Male
Age Groups: Child